CLINICAL TRIAL: NCT04552132
Title: Postoperative Pain and Healing of Molar Root Canal Teeth Using GentleWave vs. EndoActivator
Brief Title: Postoperative Pain and Healing in Teeth Treated With GentleWave or EndoActivator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, David Bingham, DDS, Endodontic Resident at the Center for Advanced Dental Education, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31359
Record Dates: First submitted 2020-09-13; First posted 2020-09-17 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Symptomatic Irreversible Pulpitis; Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GentleWave (Experimental): Patients randomly assigned to the GentleWave group will receive irrigation and activation of irrigants with the GentleWave device (multisonic energy) by Sonendo.
  Interventions: Device: Multisonic vs Sonic activation of irrigants
- EndoActivator (Active Comparator): Patients randomly assigned to the EndoActivator group will receive irrigation via a side-vented needle and activation using the EndoActivator (sonic energy) by Dentsply Sirona.
  Interventions: Device: Multisonic vs Sonic activation of irrigants

INTERVENTIONS:
Device: Multisonic vs Sonic activation of irrigants — Energy is input into the intracanal irrigants for activation in the hopes of increasing irrigant efficacy.

SUMMARY:
Patients with painful molars will be randomly assigned to 2 different groups: GentleWave and EndoActivator. The root canals will be completed using identical protocols except in the mode of delivery and activation of irrigation (using either the GentleWave or EndoActivator). Postoperative pain and pain pill consumption will be measured for the 4 days following their root canal using a Visual Analog Scale and Pain Pill Log, respectively. The alternative hypothesis is that patients undergoing treatment using the GentleWave will experience less pain postoperatively and will consume fewer pain pills.

A 12-month follow up with exam and radiographs will be completed to evaluate healing.

ELIGIBILITY:
Inclusion Criteria:

• Adults, able to provide informed consent, with restorable symptomatic molars reporting preoperative pain ≥20mm on a 100mm Visual Analog Scale (VAS) during the previous 24 hours.

Exclusion Criteria:

* Minors
* Pregnant women
* Prisoners
* Persons unable to adequately provide informed consent
* Non-restorable teeth
* Patients unable to sit in the dental chair for 3 hours
* Patients with compromised cardiac health requiring less than .08mg epinephrine
* Patients with a pacemaker
* Patients where Ibuprofen and Acetaminophen are contraindicated
* Patients unable to swallow pills
* Patients with pain originating somewhere other than the tooth in question
* Patients having taken analgesics within previous 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bingham, DDS, Principal Investigator — Resident at the Center for Advanced Dental Education; Brian Judd, DDS, Principal Investigator — Resident at the Center for Advanced Dental Education
Locations (1):
- Saint Louis University Center for Advanced Dental Education, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, no patients were excluded from the study prior to assignment of group. However, the data for one participant in the GentleWave group was excluded from final data analysis because it was determined that their preoperative pain was insufficient for the study and they should not have been enrolled in the first place.
Period: Overall Study
Arm/Group | GentleWave | EndoActivator
Started | 31 | 32
Completed | 26 | 29
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GentleWave | EndoActivator | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.33 (14.40) | 43.44 (11.98) | 43.87 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 11 | 13 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63
Pre-operative pain [Mean (Standard Deviation); unit: score on a scale] — Measured by the patient placing a mark that they feel best represents their level of pain on a 100mm Visual Analog Scale with 'No Pain' on the left (at 0) and 'Worst Pain Possible' on the right (at 100).
  score on a scale | 66.00 (24.67) | 70.80 (23.45) | 68.50 (24.15)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Postoperative Pain for Patients Seen From 09/2020-06/2021
Description: Postoperative Pain will be measured by the patient placing a mark that they feel best represents their level of pain on a 100mm Visual Analog Scale with 'No Pain' on the left (at 0) and 'Worst Pain Possible' on the right (at 100).
Time Frame: 24 hours post-operative
Population: Participants seen from 09/2020-06/2021 that completed and returned their paperwork.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 15
score on a scale | 14.75 (17.91) | 16.23 (27.93)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.63, Fisher Exact

2. Primary Outcome: 24 Hour Postoperative Pain for Patients Seen From 07/2021-03/2022
Description: as for outcome 1
Time Frame: 24 hr postoperatively
Population: Participants seen from 07/2021-03/2022 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 14 | 14
score on a scale | 12.86 (18.65) | 17.00 (18.69)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 1.00, Fisher Exact

3. Primary Outcome: 48 Hour Postoperative Pain for Patients Seen From 09/2020-06/2021
Description: as for outcome 1
Time Frame: 48 hours post-operative
Population: Participants seen from 09/2020-06/2021 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 15
score on a scale | 12.58 (18.71) | 11.73 (19.58)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.63, Fisher Exact

4. Primary Outcome: 48 Hour Postoperative Pain for Patients Seen From 07/2021-03/2022
Description: as for outcome 1
Time Frame: 48 hours post-operative
Population: Participants seen from 07/2021-03/2022 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 14 | 14
score on a scale | 6.86 (12.35) | 10.07 (11.49)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 1.00, Fisher Exact

5. Primary Outcome: 72 Hour Postoperative Pain for Patients Seen From 09/2020-06/2021
Description: as for outcome 1
Time Frame: 72 hour post-operative
Population: Participants seen from 09/2020-06/2021 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 15
score on a scale | 7.46 (14.36) | 7.30 (13.14)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.57, Fisher Exact

6. Primary Outcome: 72 Hour Postoperative Pain for Patients Seen From 07/2021-03/2022
Description: as for outcome 1
Time Frame: 72 hours post-operative
Population: Participants seen from 07/2021-03/2022 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 14 | 14
score on a scale | 3.57 (4.89) | 5.86 (10.85)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.60, Fisher Exact

7. Primary Outcome: 96 Hour Postoperative Pain for Patients Seen From 09/2020-06/2021
Description: as for outcome 1
Time Frame: 96 hours post-operative
Population: Participants seen from 09/2020-06/2021 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 15
score on a scale | 9.96 (19.98) | 7.53 (16.15)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 1.00, Fisher Exact

8. Primary Outcome: 96 Hour Postoperative Pain for Patients Seen From 07/2021-03/2022
Description: as for outcome 1
Time Frame: 96 hours post-operative
Population: Participants seen from 07/2021-03/2022 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 14 | 14
score on a scale | 1.57 (3.61) | 2.57 (3.63)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 1.00, Fisher Exact

9. Primary Outcome: Cone Beam Computed Tomography (CBCT) Healing Assessment
Description: Each tooth root was classified as healed (no periapical radiolucency), healing (periapical radiolucency educed in size), or diseased (periapical radiolucency same size or larger). Pre-operative vs. post-operative periapical health evaluated using radiographs to compare the size of periapical radiolucencies present pre-op vs post-op.
Time Frame: 12 month recall
Population: Patients that were able to return for a 12-month recall before the study ended.
Measure: Number; unit: roots
Units Other Than Participants: Roots (teeth have multiple roots)
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 14
Number analyzed (Roots (teeth have multiple roots)) | 28 | 32
roots
  Healed | 24 | 24
  Healing | 4 | 4
  Diseased | 0 | 4
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.18, Chi-squared

10. Primary Outcome: Clinical Tooth Healing Classification Based on Clinical Examination and Patient Report
Description: Teeth were classified as being clinically successful if the patient had no symptoms other than mild tenderness to percussion. Teeth were classified as failures if outside these parameters.
Time Frame: 12-month recall
Population: Patients that could return for a 12-month recall before study ended.
Measure: Number; unit: teeth
Units Other Than Participants: Teeth
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 14
Number analyzed (Teeth) | 12 | 14
teeth
  Success | 12 | 12
  Failure | 0 | 2
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = .4993, Chi-squared

11. Secondary Outcome: Pain Pill Consumption for Patients Seen From 09/2021-06/2021
Description: Patients will be given 16 tabs of 600mg Ibuprofen and 16 tabs of 650mg Acetaminophen with instructions to take 1 pill every 6 hours as needed for pain. Patients will be given a Pain Pill Log to record each time they take a pill. The total number of pills consumed will be tabulated for each patient.
Time Frame: Patient to record on the Pain Pill Log each time that they take a pain pill during the 4 days following their root canal treatment.
Population: Participants seen from 09/2020-06/2021 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 12 | 15
pills | 5.08 (4.56) | 6.63 (7.63)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = 0.52, t-test, 2 sided

12. Secondary Outcome: Pain Pill Consumption for Patients Seen From 07/2021-03/2022
Description: as for outcome 11
Time Frame: as for outcome 11
Population: Participants seen from 07/2021-03/2022 that completed and returned their paperwork
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | GentleWave | EndoActivator
Number analyzed (Participants) | 14 | 14
pills | 4.00 (3.82) | 4.93 (8.02)
Statistical Analysis 1: Comparison: GentleWave vs EndoActivator; Test type: Superiority; p = .70, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 10 months.
Arm/Group | GentleWave | EndoActivator
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04552132/Prot_SAP_000.pdf